CLINICAL TRIAL: NCT04173234
Title: The Effect on Muscle Architecture Properties and Motor Functions of Aerobic Training in Children With Duchenne Muscle Dystrophy
Brief Title: Aerobic Exercise in Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Numan Bulut, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-19022
Record Dates: First submitted 2019-05-28; First posted 2019-11-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Aerobic Training; Ultrasonography; Motor Function
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Home exercise program Children will be given a home program including stretching, breathing, normal joint movement, body weight and mildly resistant exercises, and children will be asked to do these for 3 to 5 days a week. Also, aerobic training will be performed 3 days a week for 12 weeks at 60% of their maximum hearth rate with 50 minutes total duration consisting of 10 min warm up and 10 min cool down period to children in treatment group.
  Interventions: Other: Aerobic Training; Other: Home exercise program
- Control Group (Active Comparator): Home exercise program Children will be given a home program including stretching, breathing, normal joint movement, body weight and mildly resistant exercises, and children will be asked to do this program for 5 days a week.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Aerobic Training — Aerobic training will be performed 3 days a week for 12 weeks at 60% of their maximum hearth rate with 50 minutes total duration consisting of 10 min warm up and 10 min cool down period to children in treatment group.
  Arms: Treatment Group
Other: Home exercise program — Children will be given a home program including stretching, breathing, normal joint movement, body weight and mildly resistant exercises, and children will be asked to do these for 3 to 5 days a week.

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is the most common neuromuscular disease in childhood with an estimate incidence of 1 in 3500 to 5000 male births. The effect of aerobic training on muscle architectural properties and motor functions such as muscle activation is not clear in DMD. The aim of this study is to investigate the effects of aerobic training on these parameters in children with DMD. Twenty children with DMD included in the study will be divided into two groups as home program and home program+aerobic training with block randomization method. Home program including stretching, respiratory, range of motion and mild resistance exercise with body weight will be asked to apply 3-5 days a week for 12 weeks, aerobic training will be performed 3 days a week for 12 weeks at 60% of their maximum hearth rate with 50 minutes total duration consisting of 10 min warm up and 10 min cool down period. Muscle architectural properties, muscle strength, muscle activation and motor function will be assessed with ultrasonographic, hand-held myometry, surface EMG and Motor Function Measure, consecutively. Assessments will be applied at pre-training and after 12 weeks of training.

ELIGIBILITY:
Inclusion criteria:

* Children had diagnosis of DMD confirmed by genetic analysis,
* Children had functional level of Grade 1 and 2 according to Vignos Scale.

Exclusion criteria:

* Children had undergone any surgery or suffered injury of the lower limbs,
* Children had comorbid disease
* Children were applied regular aerobic training in last 6 months.

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Because DMD is X linked recessive disorder, this disorder is seen in male.
Enrollment: 19 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Muscle Thickness, Fascicle Length, Pennation Angle with Ultrasonography | 10 minutes
  Bilateral Vastus Lateralis and Medial Gastrocnemius US evaluations were performed with use of a 5-10 MHz linear probe (Diasus Dynamic Imaging Ltd, Livingston, Scotland,UK). Children were positioned supine with their legs extended and their muscles relaxed for vastus lateralis.Children were positioned prone position with their legs and their muscles relaxed for medial gastrocnemius. While Muscle Thickness and Fascicle Length would be expressed as centimeters, pennation angle would be angularly indicated.

SECONDARY OUTCOMES:
Assessment of Motor Function by Motor Function Measure (MFM) | 30 minutes
  The total scores of the MFM test were determined in three motor function domains: D1 (Standing Position & Transfers), D2 (Axial and Proximal Motor Function) and D3 (Distal Motor Function) (scored between 0-96 points, low score indicate low performance.)
Evaluation Motor Performance with Timed Functional Test and Six minute walk test | 20 minutes
  Timed function tests included time taken to stand from a supine position, time taken to run/walk 10 m, time taken to climb 4 standard-sized stairs, time taken to descend 4 standard-sized stairs and time taken to stand one leg stance (both leg).Participants were instructed to travel as far and as fast as possible in six minutes on 25 meter-indoor course.
Shortening assessment of trunk and lower extremity muscles with goniometric measurement and tape | 20 minutes
  Assessment of back extensors, hip flexors, hamstring, quadriceps and gastrocnemius muscles. For assessment back extensors, The child was placed in the supine position with his knee fixed at a neutral position, and then shortening was evaluated by having bilateral hip flexion made. For hip flexor, The child was placed in the supine position with his knee fixed at a neutral position, and he was then evaluated by having one leg hip flexion made. Hamstring shortening was measured in a supine position with the hip flexed at 90° and the opposite knee and hip were placed in an extended position. Quadriceps shortening was assessed in a prone position and then by bending knee. For gastrocnemius muscle, the child was placed in a supine position and asked to perform passive ankle dorsiflexion while the knee was extended.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No